CLINICAL TRIAL: NCT00671177
Title: Clinical Evaluation of Water Immersion Colonoscopy Insertion Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roy Soetikno, Clinical Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Protocol10642
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Colonoscopy; Digestive System; Endoscopy; Gastrointestinal Disease
Keywords: colonoscopy; diagnostic techniques; digestive system; endoscopy; gastrointestinal
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Water Immersion Colonoscopy (Experimental): Water Immersion Colonoscopy
  Interventions: Procedure: water immersion colonoscopy
- Standard Air Colonoscopy (Active Comparator): Standard Air Colonoscopy
  Interventions: Procedure: standard air colonoscopy

INTERVENTIONS:
Procedure: water immersion colonoscopy — instillation of 300cc of water in the rectum
  Arms: Water Immersion Colonoscopy
Procedure: standard air colonoscopy — air instillation in colon for visualization
  Arms: Standard Air Colonoscopy

SUMMARY:
Recent studies indicate that infusing 300 milliliters of water (in lieu of air) into the rectum and left colon through the colonoscope as it is being inserted during a colonoscopy examination can allow easier endoscope advancement. This method may prevent stretching of the colon, and ultimately reduce pain induced during colonoscopy. Improvements in patient comfort and cooperation, may increase the efficiency and success rate of complete colonoscopy. The purpose of the study is to test the efficacy of the water immersion technique in patients colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* presentation for colonoscopy
* male
* age 18 or older

Exclusion Criteria:

* women
* known inflammatory bowel disease
* presentation for emergency colonoscopy
* history of partial colectomy
* chronic narcotic or benzodiazepine use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Soetikno, MD, MS, Principal Investigator — VA Palo Alto/Stanford University Medical Center
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung CW, Kaltenbach T, Soetikno R, Wu KK, Leung FW, Friedland S. Water immersion versus standard colonoscopy insertion technique: randomized trial shows promise for minimal sedation. Endoscopy. 2010 Jul;42(7):557-63. doi: 10.1055/s-0029-1244231. Epub 2010 Jun 30. PMID 20593332

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Water Immersion Colonoscopy | Standard Air Colonoscopy
Started | 114 | 115
Completed | 112 | 114
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water Immersion Colonoscopy | Standard Air Colonoscopy | Total
Number analyzed (Participants) | 112 | 114 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.9) | 62.5 (8.9) | 62.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 112 | 114 | 226

OUTCOME MEASURES:

1. Primary Outcome: Colonoscopy Success With Minimal Sedation
Time Frame: At the time of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Water Immersion Colonoscopy | Standard Air Colonoscopy
Number analyzed (Participants) | 112 | 114
Participants | 57 | 32

2. Secondary Outcome: Time to Cecum
Time Frame: At the time of the procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Water Immersion Colonoscopy | Standard Air Colonoscopy
Number analyzed (Participants) | 112 | 114
minutes
  Attending | 5.4 (5.9) | 7.2 (5.8)
  Trainee | 13 (7.5) | 20.5 (13.9)

3. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction was measured on a scale of 1 (best) to 7 (worst).
Time Frame: At the time of the procedure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Water Immersion Colonoscopy | Standard Air Colonoscopy
Number analyzed (Participants) | 112 | 114
units on a scale | 1.09 [1 to 7] | 1.26 [1 to 7]

ADVERSE EVENTS:
Arm/Group | Water Immersion Colonoscopy | Standard Air Colonoscopy
Serious Adverse Events (participants affected / at risk) | 0/1114 | 0/115
Other Adverse Events (participants affected / at risk) | 0/114 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No